CLINICAL TRIAL: NCT01405612
Title: An Open-label, Single Centre, Randomised, Cross-over Study to Examine the Effect of Ulimorelin on the Pharmacokinetics of Midazolam After Repeat Dose Administration of Ulimorelin in Healthy Volunteers
Brief Title: Study to Examine the Effect of Ulimorelin on the Pharmacokinetics of Midazolam in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NPJ5004-02/2011 (DDI)
Record Dates: First submitted 2011-07-22; First posted 2011-07-29 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Digestive System Disorders
MeSH Terms: conditions — Digestive System Diseases | interventions — Midazolam; ulimorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Experimental): Those subjects to receive Treatment A will receive a single dose of midazolam on Day 1 and will be discharged from the study unit on Day 2, at least 30 hours after midazolam dosing.
  Interventions: Drug: Midazolam
- Ulimorelin (Experimental): Those subjects to receive Treatment B will receive once daily ulimorelin on Days 1 to 5. Midazolam will be administered on Day 5 with the last dose of ulimorelin and subjects will be discharged from the study unit on Day 6, at least 30 hours after midazolam dosing.
  Interventions: Drug: Ulimorelin

INTERVENTIONS:
Drug: Midazolam — Single oral administration on Day 1 or Day 5
  Arms: Midazolam
Drug: Ulimorelin — Intravenous infusion of 480 micrograms/kg on Days 1 to 5
  Other Names: TZP101
  Arms: Ulimorelin

SUMMARY:
An open-label, single centre, randomised, cross-over study to examine the effect of ulimorelin on the pharmacokinetics of midazolam after repeat dose administration of ulimorelin in healthy volunteers.

DETAILED DESCRIPTION:
Ulimorelin is a first-in-class new chemical entity. It is a ghrelin agonist with gastroprokinetic activity being developed as an intravenous therapy to be used in the treatment of gastrointestinal (GI) hypomotility disorders such as post-operative ileus (POI) and gastroparesis.

POI is a transient disruption of co-ordinated bowel motility that contributes to patient morbidity, discomfort and prolonged recovery times. POI most commonly occurs after abdominal surgery and annually, POI is the main determinant of length of hospital stay after major abdominal surgery and a factor in patient hospital re-admissions, increased healthcare resource use and cost, and decreased patient satisfaction. Current strategies to attenuate POI are aimed at enhanced recovery after surgery (ERAS) or "fast track". These are multimodal care protocols designed to reduce the impact of external and internal factors on POI duration. Recently, fewer complications and a quicker return to work and normal activities for patients who have had ERAS programmes implemented have been reported. In spite of these strategies only up to 20% of subjects undergoing partial bowel resection recover GI function within 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers (as determined by medical history, physical examination, laboratory test values, vital signs and 12-lead ECGs at screening) aged 18 to 45 years.
2. Non-smokers from three months before receiving the first dose of study drug and for the duration of the study.
3. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
4. Body weight ≥ 50 kg and ≤ 120 kg at screening.
5. Able to voluntarily provide written informed consent to participate in the study.
6. Must understand the purposes and risks of the study and agree to follow the restrictions and schedule of procedures as defined in the protocol, as confirmed during the informed consent process.
7. Female volunteers must be postmenopausal (for at least one year and confirmed by serum follicle stimulating hormone (FSH) at screening), surgically sterile, practising true sexual abstinence, or must use two highly effective methods of contraception (defined as a failure rate of less than 1% per year when used consistently and correctly) throughout the study until after post-study medical as follows: contraceptive implants, injectables, oral contraceptives, some intrauterine devices (IUDs), vasectomised partner and / or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository.
8. Hormonal and IUD methods of contraception must be established for a period of three months prior to dosing and cannot be changed or altered during the study.
9. Females of childbearing potential must have a negative serum pregnancy test at screening (β-hCG) and a negative urine pregnancy test at check-in for each period.
10. Sexually active male volunteers must use condoms with their partners throughout the study and for 90 days after completion of the study in addition to their partner's normal mode of contraception.
11. Male volunteers must not donate sperm during the study and for 90 days after completion of the study.
12. Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).
13. The volunteer's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical study.

Exclusion Criteria:

1. Subjects with history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or current infection.
2. Pregnant or lactating females.
3. Laboratory values at screening which are deemed to be clinically significant, unless agreed in advance by the Sponsor's Medical Representative and Principal Investigator, or a value of alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than 10% of the upper limit of the reference range.
4. Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
5. Current or history of drug or alcohol abuse or a positive drugs of abuse test at screening or check-in.
6. Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
7. Any significant illness during the screening period preceding entry into this study.
8. Donation of blood or blood products within 90 days prior to study drug administration, or at any time during the study, except as required by this protocol or haemoglobin < 12.0 g/dl at screening.
9. Subjects who have received monoamine oxidase inhibitors or who have been on a special diet as assessed by the Investigator within 28 days of starting the study or during the study.
10. Subjects who have a history or presence of any significant drug allergy, or a known allergy or contraindication to midazolam or other benzodiazepines.
11. Use of any prescription or over-the-counter medication (including vitamins, herbal and mineral supplements) within 28 days prior to study drug administration until the end of the study, with the exception of Investigator-approved hormonal contraceptives, hormone replacement therapy (HRT) and occasional paracetamol.
12. Use of any known inhibitors or inducers (e.g. St. John's Wort) of CYP3A4 within 28 days or 5 half lives prior to study drug administration, whichever is longer, until the end of the study.
13. Use of grapefruit juice or grapefruit containing products within 7 days prior to study drug administration until the end of the study.
14. Strenuous exercise, as judged by the Investigator, within 72 hours prior to screening, within 72 hours prior to study drug administration and for the duration of the study (until post-study medical).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
AUC(0 to infinity) of midazolam | Pre-(midazolam)dose and 15, 30, 45 mins and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 30 hours post dose
Cmax of Midazolam | Pre-(midazolam)dose and 15, 30, 45 mins and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 30 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tomas, PhD, Study Director — Norgine
Locations (1):
- BioKinetic Europe Ltd, Belfast, United Kingdom